CLINICAL TRIAL: NCT05460442
Title: Comparison of Ultrasound-Guided Pericapsular Nerve Group Block Versus Ultrasound-Guided Fascia Iliaca Block for Pediatric Hip Surgery
Brief Title: Pericapsular Nerve Group Block Versus Fascia Iliaca Block for Pediatric Hip Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Elsaied Mohamed Hosny Alam, Resident of Anesthesiology and Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 35436/4/22
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Hip Surgery; Pericapsular Nerve; Fascia Iliaca

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caudal Block group (Experimental): 25 patients will receive ultrasound-guided caudal block with bupivacaine 0.25% (0.5 mL/kg) after induction of anesthesia.
  Interventions: Procedure: Caudal Block group
- Pericapsular nerve group block (Experimental): 25 patients will receive ipsilateral ultrasound-guided Pericapsular nerve group block with bupivacaine 0.25% (0.5 mL/kg) after induction of anesthesia.
  Interventions: Procedure: Pericapsular nerve group block
- Fascia iliaca group (Experimental): 25 patients will receive ipsilateral ultrasound-guided Fascia iliaca compartment block with bupivacaine 0.25% (0.5 m. L/kg) after induction of anesthesia.
  Interventions: Procedure: Fascia iliaca group

INTERVENTIONS:
Procedure: Caudal Block group — Patients will be placed in the lateral decubitus position. After local sterilization with povidone-iodine, the sacral hiatus will be visualized at the level of the sacral Cornus by ultrasound. The needle will be advanced toward the upper third of the sacrococcygeal ligament. The needle advancement will be terminated immediately after penetrating the sacrococcygeal ligament. At this level, after confirming the absence of blood or cerebrospinal fluid on aspiration, bupivacaine 0.25% (0.5 mL/kg) will be injected over 1 minute
  Arms: Caudal Block group
Procedure: Pericapsular nerve group block — Patients will receive ultrasound-guided Pericapsular nerve group block in the supine position after proper sterilization of the groin region. The needle will be inserted in-plane with the transducer. The Pericapsular nerve group block group will receive 0.5 mL/kg of (0.25%) bupivacaine after a negative aspiration
  Arms: Pericapsular nerve group block
Procedure: Fascia iliaca group — Patients will receive Ultrasound-Guided fascia iliaca compartment block in the supine position after sterilization of groin area. The needle will be inserted in-plane with the transducer. The needle tip will be advanced through the fascia iliaca and inserted further cephalad just below the fascia iliaca into the iliacus muscle. 0.5 mL/kg of (0.25%) bupivacaine will be injected and visualized moving cephalad away from the needle tip
  Arms: Fascia iliaca group

SUMMARY:
This compares the postoperative analgesic effect of ultrasound-guided pericapsular nerve group block (PENG) with ultrasound-guided fascia iliaca compartment block in pediatric patients undergoing hip surgery.

DETAILED DESCRIPTION:
Surgeries involving hip joints in pediatric patients are associated with severe intraoperative and postoperative pain despite the use of systemic opioids.

Caudal block is the most commonly used method of regional anesthesia in children to control intraoperative and postoperative pain in surgeries involving lower limbs. However, there have been many side effects of caudal block such as hypotension, urine retention, excessive motor block, technical failure, nausea, and vomiting which may limit its use.

There are several techniques of ultrasound-guided regional anesthesia that are used to control acute pain in hip surgery with fewer side effects such as a lumbar plexus block, femoral nerve block, or a fascia iliaca compartment block.

The fascia iliaca compartment block (FICB) was described in 1989. It remains a popular regional anesthetic technique for surgical procedures involving the hip joint and femur. Local anesthetic (LA) is injected proximally beneath the fascia iliaca to block the femoral nerve (FN), obturator nerve (ON), and lateral cutaneous nerve of the thigh (LCNT) simultaneously.

The pericapsular nerve group (PENG) block was introduced to block the articular branches of the femoral, obturator, and accessory obturator nerves which provide sensory innervation to the hip. This regional anesthetic technique was described in 2018 for acute analgesia related to hip fractures.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients
* aged 1-6 years old
* both sexes,
* American Society of Anesthesiologists (ASA) physical activity class I-II
* scheduled for elective hip surgery under general anesthesia.

Exclusion Criteria:

* Children with the severe systemic disease with American Society of Anesthesiologists physical activity class III or IV.
* Children with previous neurological or spinal disorders.
* Coagulation disorder.
* Infection at the block injection site.
* History of allergy to local anesthetics.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-07-20 (Estimated); Study Completion 2023-07-29 (Estimated)

PRIMARY OUTCOMES:
Total Opioids consumption | 24 hours postoperatively
  Total Opioids consumption in first 24 hour postoperatively will be recorded

SECONDARY OUTCOMES:
Postoperative pain | At post anesthesia care unit then after 30 minutes 2, 4, 6, 12, 24 hours.
  Postoperative pain which will be assessed by face, legs, activity, and cry consolability scale [FLACC]
Time to first rescue analgesia | 24 hours Postoperatively
  Time of administration of first rescue analgesia will be recorded.
Adverse effects | 24 hours Postoperatively
  Adverse effects: hypotension, Bradycardia, hematoma, and local anesthetic toxicity will be observed and treated accordingly.
Heart rate | Intraoperative then at post anesthesia care unit then after 30 minutes 2, 4, 6, 12, 24 hours
  Perioperative heart rate will be observed
Mean arterial blood pressure | Intraoperative then at post anesthesia care unit then after 30 minutes 2, 4, 6, 12, 24 hours.
  Perioperative mean arterial blood pressure will be observed

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available under a reasonable request from the corresponding author
Supporting Information: Study Protocol
Time Frame: One year after the end of the study